CLINICAL TRIAL: NCT05909306
Title: Development of a Partograph E-learning Tool and Evaluation of Its Efficiency in Student Midwives in Turkey: A Randomized Controlled Experimental Study
Brief Title: Development of a Partograph E-learning Tool and Evaluation of Its Efficiency in Student Midwives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Damla Kizilca Cakaloz, Research Assistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Interventional study in Turkey
Record Dates: First submitted 2023-06-12; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Midwifery Students Education
Keywords: Partograph; e-learning; midwifery; e-partograph

STUDY DESIGN:
Intervention Model Description: The complete randomization technique was used to assign students to groups. Following recruitment, the midwifery students were divided into an education and a control group by randomization. The first half of the list consisting of numbers produced randomly showed the students to be assigned to the education group and the other half indicated the students to be assigned to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): The education group was applied partograph education in addition to formal education by using the partograph e-learning tool that was developed.
  Interventions: Other: Education Group
- Control Group (No Intervention): The control group continued their formal education.

INTERVENTIONS:
Other: Education Group — Two online meetings were planned with the education group. In the first meeting, an average of 35-minute-long live lecturing was performed on filling out the data forms and using the partograph e-learning tool through e-learning tool created in the first interview. The researcher held the second interview one week after the first one. In the second interview, a live lecture lasting 30 minutes was given to talk about and solve the problems that students experienced with the partograph e-learning tool and answer the questions. The partograph e-learning tool was kept open for one month for the students in the education group. At the end of the one-month education, the students were asked to fill out the post-test (Academic Achievement Test) defined in the system. After the post-test was completed, the system was closed to the access of the students in the education group and made available to the students in the control group.
  Arms: Education Group

SUMMARY:
A randomized control trial was made to develop a partograph e-learning tool and evaluate its effectiveness in student midwives in Turkey.

DETAILED DESCRIPTION:
With the use of a partograph, complications are detected and intervened promptly, and unnecessary applications are avoided. Therefore, it has become an integral part of the practices of midwives who manage normal births under their responsibility to reduce maternal and neonatal morbidity and mortality. One of the intrapartum care services of midwives is to detect prolonged labor, especially with the use of a partograph, and to apply quick and accurate intervention. However, the partograph is not widely used all over the world at the desired level.

Recently, the use of the e-learning system, which is recommended as a method of obtaining and perceiving information easily, has increased considerably. Although this is a new concept in our country, it has started to be adopted rapidly.

In our country, there is no study on the use of e-learning in midwifery practices. However, in many international studies, it is stated that e-learning is acceptable and more practical and effective than classical methods in midwifery education and practices. This research was designed as a randomized controlled experimental study to develop an e-learning tool that could be an alternative to midwifery students' learning of the use of a partograph and to evaluate its effectiveness.

The hypothesis was tested that there is a significant difference between the students who received and did not receive training with the partograph e-learning tool in terms of post-test education achievement scores. In addition, it was found that there is a significant difference between the pre-test and post-test education achievement scores of the students who received training with the partograph e-learning tool.

ELIGIBILITY:
Inclusion Criteria:

* Studying in the 3rd year of the midwifery undergraduate program
* Those who took the Childbirth and Postpartum Period Lecture and enrolled in the Childbirth and Postpartum Period At Risk Lecture
* Able to use the internet and computer
* Having an e-mail address with which he can communicate over the internet
* Students with internet access

Exclusion Criteria:

* Students who could not continue their education due to reasons (Registration freeze, lateral transfer, health problems, etc.) were excluded from the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Acadeic Achievement Test before intervention (Pretest) | After randomization, in the first meeting
  The Academic Achievement Test consisted of eight multiple-choice questions and two case scenarios about knowledge, skills, and synthesis on the use of the partograph in labor. For each question regarding the partograph knowledge level, correct answers were scored 2 and incorrect answers 0. The minimum score on the knowledge is a 0; maximum is 16. For partograph filling skills, students systematically reviewed each case and filled out partographs with the given information and were evaluated one by one according to individual partograph components. The minimum score on the both cases are a 0; maximum is 34. For the partograph synthesis, open-ended interpretation questions were added to the end of each case. The minimum score on the partograph synthesis are a 0; maximum is 10. In total, the minimum possible score on the the Academic Achievement Test is a 0; maximum is 60. Higher scores indicate greater levels of Academic Achievement.
Acadeic Achievement Test after intervention (Posttest ) | One month after the pretest.
  The Academic Achievement Test consisted of eight multiple-choice questions and two case scenarios about knowledge, skills, and synthesis on the use of the partograph in labor. For each question regarding the partograph knowledge level, correct answers were scored 2 and incorrect answers 0. The minimum score on the knowledge is a 0; maximum is 16. For partograph filling skills, students systematically reviewed each case and filled out partographs with the given information and were evaluated one by one according to individual partograph components. The minimum score on the both cases are a 0; maximum is 34. For the partograph synthesis, open-ended interpretation questions were added to the end of each case. The minimum score on the partograph synthesis are a 0; maximum is 10. In total, the minimum possible score on the the Academic Achievement Test is a 0; maximum is 60. Higher scores indicate greater levels of Academic Achievement.

CONTACTS AND LOCATIONS:
Overall Officials: Damla Kizilca Cakaloz, PhD, Study Chair — Adnan Menderes University, Faculty of Health Sciences, Division of Midwifery; Ayden Coban, PhD, Study Director — Adnan Menderes University, Faculty of Health Sciences, Division of Midwifery
Locations (1):
- Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.